CLINICAL TRIAL: NCT03343561
Title: Effect of Dietary Intervention on Gut Microbiome in Hong Kong Obese Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Prenetics Limited (Unknown)
Responsible Party: Principal Investigator, Prof. Man-sau WONG, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FSTRC2017PIS
Record Dates: First submitted 2017-11-01; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: As soon as the samples are obtained from the subjects, subjects will be coded straight-away. No samples will be stored with the subjects' name on, only codes will be used. Only the investigating team will be able to break the codes and trace the results back to the subjects. All the questionnaires will be only shown the subjects' code without subjects' name on them. No data file in hard or soft copy format will contain all the information on the subject's name, project code and experiment result.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Subjects would have subjects' own diet as usual
- Intervention diet 1 (Experimental): Nutrition advice will be given to subjects to consume a healthy diet and select food with Polyunsaturated fatty acids like fish and nuts to replace subjects' own food in high fat
  Interventions: Behavioral: Nutrition Advice
- Intervention diet 2 (Experimental): Nutrition advice will be given to subjects to consume a healthy diet and select food with whole grains to replace subjects own food in carbohydrate
  Interventions: Behavioral: Nutrition Advice
- Intervention diet 3 (Experimental): Nutrition advice will be given to subjects to consume a healthy diet and select food with healthy choices in fat and carbohydrate to replace subjects' own food choice
  Interventions: Behavioral: Nutrition Advice

INTERVENTIONS:
Behavioral: Nutrition Advice — Intervention diet for 8 weeks for intervention group. Detailed 30 mins consultation in week 1 (provided by dietitian) and 15 min consultation (provided by RA) in week 4 to enhance subject adherence to the diet for intervention group. Control group subjects will receive 1 detailed 30 mins nutrition consultation from dietitian after the study.
  Arms: Intervention diet 1; Intervention diet 2; Intervention diet 3

SUMMARY:
Modern way of life characterized by decreased physical activity and poor dietary habits seems to be an important trigger for the onset of metabolic disorders. Accumulating evidence indicates that the gut microbiota is involved in host metabolism by increasing energy extraction, immune system modulation, and altering lipid metabolism, which play an intricate role in metabolic disorders, such as obesity and diabetes. Diet has a major role in shaping the composition and activity of gut microbiota. Consumptions of whole-grain and polyunsaturated fatty acids are known to exert certain extent of impacts on gut microbial communities in terms of participants' richness and diversity. In this study, the investigators aim to evaluate the impact of dietary intervention on gut microbiome in Hong Kong obese population

DETAILED DESCRIPTION:
1. Purpose of the Study Modern way of life characterized by decreased physical activity and poor dietary habits seems to be an important trigger for the onset of metabolic disorders. Accumulating evidence indicates that the gut microbiota is involved in host metabolism by increasing energy extraction, immune system modulation, and altering lipid metabolism, which play an intricate role in metabolic disorders, such as obesity and diabetes. Diet has a major role in shaping the composition and activity of gut microbiota. Consumptions of whole-grain and polyunsaturated fatty acids are known to exert certain extent of impacts on gut microbial communities in terms of the participants' richness and diversity. In this study, the investigators aim to evaluate the impact of dietary intervention on gut microbiome in Hong Kong obese population.
2. Method of investigation

   The study will last for 9 weeks. 48 eligible subjects aged 30-60 years old will be randomly allocated into 4 groups, to 3 of which nutrition advice on healthy diets and preferred food choices will be given while the remaining one will keep the participants' usual diets. Dietary surveys will be conducted to reveal the participants' dietary habits. Meanwhile, blood, stool and buccal swab will be collected to examine the effect of dietary intervention for example, changes of composition of gut microbiota, fasting blood glucose levels and lipid profiles as well as other metabolic indicators.
3. Approach

Subjects will be recruited via convenience sampling through internet and poster promotion. Screening for eligible subjects will be conducted by Research staff in PolyU on phone. If the participants are interested to join the study, the staff will explain study details and appointments will thus be made on a first come first serve basis. The study starts upon obtained consensus from subjects. Blood collection and testing will be outsourced to health check centre to further confirm the eligibility of subjects.

Eligible subjects will be randomly allocated into either control or intervention groups, in which subjects will receive dietitian consultations provided by registered dietitians. Also, stool, blood and buccal swab samples of subjects will be collected at various time points to examine changes of the investigators' desired parameters within the study.

ELIGIBILITY:
Inclusion Criteria:

* With BMI >23kg/m2 Asian subjects, aged 30-60 years old

Exclusion Criteria:

* Chronic, clinically significant (unresolved, requiring on-going medical management or medication) pulmonary, cardiovascular (e.g. heart disease, high blood pressure etc.), gastrointestinal, hepatic or renal functional abnormality, and metabolic syndrome as determined by medical history or physical examination.
* History of active uncontrolled gastrointestinal disorders or diseases including: inflammatory bowel disease (IBD) including ulcerative colitis (mild-moderate-severe), Crohn's disease (mild-moderate-severe), or indeterminate colitis; irritable bowel syndrome (IBW) (moderate-severe); persistent, infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhea of unknown etiology, Clostridium difficile infection (recurrent) or Helicobacter pylori infection (untreated); chronic constipation
* Major surgery of the GI tract, with the exception of cholecystectomy and appendectomy, in the past five years. Any major bowel resection at any time.
* Use of any of the following drugs within the 1 months sampling: systemic antibiotics, (intravenous, intramuscular, or oral); oral, intravenous, intramuscular, nasal or inhaled corticosteroids; cytokines; methotrexate or immunosuppressive cytotoxic agents; large doses of commercial probiotics consumed (greater than or equal to 108 cfu or organisms per day) - includes tablets, capsules, lozenges, chewing gum or powders in which probiotic is a primary component. Ordinary dietary components such as fermented beverages/milks, yogurts, foods do not apply.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — M:F ratio is 1:1
Enrollment: 48 (Estimated)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbial Abundance Profile using QIIME 2.0 | 6 months
  Microbial Abundance Profile is a commonly used metric to assess the impact of interventions on microbial community (References: 1. The Human Microbiome Project Consortium. A framework for human microbiome research. Nature 486, 215-221 (2012). 2. Wu et al. Linking Long-Term Dietary Patterns with Gut Microbial Enterotypes. Science. 2011 Oct 7; 334(6052): 105-108;)

CONTACTS AND LOCATIONS:
Overall Officials: Man-sau WONG, Doctoral, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This study has registered in the system of clinical trial in HKU — http://www.hkuctr.com/Study/Print/7254f25c576d4e0da87678892275247d